CLINICAL TRIAL: NCT06376461
Title: Prospective, Multicentre Study to Validate the GastroIntestinal Dysfunction Score (GIDS) and Describe Prevalence, Outcomes, and Management of Phosphate Disorders in Intensive Care Patients
Acronym: GUTPHOS
Status: Completed | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 333874
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Dysfunction
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Sites will recruit all consecutive adult patients admitted to ICU, to a maximum of 120 patients or a maximum recruitment period of 8 weeks, whichever comes first

SUMMARY:
Part A Multiple organ dysfunction syndrome is one of the main problems in critically ill patients. Several organ dysfunctions are routinely and systematically monitored in patients admitted to intensive care units. Gastrointestinal dysfunction is currently not included in multiple organ dysfunction scores and lacks a standardised approach. At the same time, investigators earlier studies have shown that gastrointestinal dysfunction plays an essential role in the course of illness in intensive care patients. A tool for measuring dysfunction is needed to enable future studies on interventions to improve gastrointestinal function. The GIDS (GastroIntestinal Dysfunction Score) combines different clinical signs and symptoms commonly observed and documented in patients in the ICU into a scoring system, allowing distinguishing between different grades of severity of dysfunction. The investigators will only use observations documented during the patient's stay in the intensive care unit without additional measurements and calculate gastrointestinal (GIDS) and other organ dysfunction scores.

Part B Phosphate is an electrolyte commonly measured and often corrected, while the indications and clear guidance for correction are insufficiently studied. The results of this study will assist in specifying indications for the correction of phosphate levels better and refine the management strategies in the future. Only phosphate levels measured as part of routine care will be documented, no additional samples for study purposes will be taken, and the study will not influence the treatment of phosphate disorders.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU during the study period (the patients already in the ICU at the time the study starts will not be included);
* Age ≥18 years;
* In participating centres in part B, serum Pi should be measured daily.

Exclusion Criteria:

* Age <18 years;
* Patients with restrictions of care such as "no intubation" or "no RRT" on ICU admission and patients admitted for treatment as organ donors;
* Continuous chronic home ventilation for neuromuscular disease;
* Declined participation or informed consent (if the local ethics committee requests the latter for this non-interventional study);
* Readmission to ICU during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU within in the recruitment period will be recruited to the trial.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
28 day outcome | 28 days after ICU admission
  28 day all cause mortality
90 day outcome | 90 days after ICU admission
  90 day all cause mortality

SECONDARY OUTCOMES:
ICU length of stay | 28 days after admission to ICU
  ICU length of stay/days alive and free of ICU by day 28
ICU length of stay | 90 days after admission to ICU
  ICU length of stay/days alive and free of ICU by day 90
Hospital length of stay | 28 days after admission
  Hospital length of stay/days alive and free of hospital by day 28
Hospital length of stay | 90 days after admission
  Hospital length of stay/days alive and free of hospital by day 90
Free of organ support | 28 days after admission
  Days alive and free of organ support (including PN free days) by day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No